CLINICAL TRIAL: NCT05266118
Title: Patient Reported Symptoms the First Week After Intensive Care Unit Discharge and up to Hospital Discharge
Status: Completed | Type: Observational
Sponsor: Ostfold Hospital Trust (Other)
Collaborators: Norwegian Nurses Organisation (Other)
Responsible Party: Sponsor
Other Study IDs: 361816
Record Dates: First submitted 2022-01-21; First posted 2022-03-04 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2022-02

CONDITIONS: Symptoms and Signs; Symptom Cluster; Follow-up Care; Critical Illness
Keywords: Critical ill; PICS; Ward; Follow-up care; Symptoms and Signs
MeSH Terms: conditions — Signs and Symptoms; Syndrome; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Former ICU patients: Participants is former ICU patients, immediately after transferred from ICU to a hospital ward. At least one of these criteria is needed for the participation in the study: ICU stays > 24 hours; ventilatory support; transferals to other ICU < 24 hours; continuous infusion of vasoactive substances. In addition, to be included, the patients must be more than 18 years of age; understand and be able to write and read Norwegian; be able to communicate verbally; not have a manifest cognitive deficit; and not being readmitted to ICU < 72 hours

SUMMARY:
The overall objective of this study is a) to increase knowledge about ICU patient's symptoms and symptom clusters during the first week after ICU discharge, and b) to identify cognitive, psychological, and physical symptoms and health state at hospital discharge.

DETAILED DESCRIPTION:
Several studies have examined how ICU patients experience being in the ICU, and up to 75% of ICU patients experience multiple intensive care related symptoms while in the ICU. Other studies have examined ICU patients' transfer from ICU to hospital wards, and the transfer may cause mixed emotions for the patient, both positive perception of an improvement in the patient's condition, but also negative perception of decreased monitoring of the patient and less staff involvement in their care. Further, extensive literature exists examining the long-term effects of being an ICU patient, and a major proportion of ICU survivors develop a combination of cognitive, psychological, and physical symptoms, which can persist for months or even years after hospital discharge. This phenomena is now recognized as post intensive care syndrome (PICS). These consequences are associated with a combination of reduced quality of life, impaired functional status and impaired daily functioning, and has consequences for both ICU survivors and their families. However, studies about what ICU patients' experience just after ICU discharge (in hospital wards), is scarce. In this time, patients are still in need of advanced personalized care after having survived critical illness and intensive care treatment.

This study will increase knowledge about symptoms and symptom clusters in ICU patients during the first week after ICU discharge, and at hospital discharge. In these areas, evidence is lacking. This knowledge will help health care providers to optimize and improve patient care and recovery during the first time period after critically illness, by providing more tailored symptom management at the right time in future support strategies and future plans for rehabilitation.

The present study is a single-center study and has a prospective, longitudinal design. A set of different symptoms are measured in 170 former ICU patients the first week after ICU discharge, in addition to a set of cognitive, psychological, and physical symptoms and health state at hospital discharge. We will measure:

1. Totally 32 different symptoms on day 1; day 3; day 5; and day 7 after ICU discharge
2. A set of cognitive (assessing the level of cognitive function), psychological (posttraumatic stress, anxiety, depression), and physical symptoms (activities of daily life) and health status at hospital discharge. The same set of questionnaires will be filled in during ward stay reflecting patient situation one week prior to ICU admittance (used as baseline measures).

ELIGIBILITY:
Inclusion criteria: Participants is former ICU patients over 18 years, immediately after transferred from ICU to a hospital ward

At least one of these criteria is needed for the participation in the study:

* ICU stays > 24 hours
* Ventilatory support
* Transferals to other ICU < 24 hours
* Continuous infusion of vasoactive substances

Exclusion criteria:

* Not able to understand, read or write Norwegian
* Not able to communicate verbally
* A manifest cognitive deficit (e.g., dementia or delirium)
* Re-admission to ICU < 72 timer

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The target group of this study is former ICU patients. The patients will be recruited from a hospital in the South-Eastern part of Norway. In this hospital, ICU patients are treated in two different ICUs, one eight-bed mixed medical/surgical ICU (treating patients with both non-invasive and invasive mechanical ventilation) and one ten-bed medical ICU (treating patients with non-invasive ventilation only). The hospital wards may be both surgical and medical wards.
Sampling Method: Probability Sample
Enrollment: 177 (Actual)
Dates: Start 2022-04-19 (Actual); Primary Completion 2022-12-21 (Actual); Study Completion 2023-03-02 (Actual)

PRIMARY OUTCOMES:
Multiple symptoms | Up to 1 week after ICU discharge
  Multiple symptoms is measured with the Memorial Symptoms Assessment Scale (MSAS).The patients will be asked to indicate whether they experience 32 different symptoms (i.e., occurence). Those who experience a symptom will be asked to rate its frequency (from rarely [1 point] to almost constantly [4 points]); intensity (from slight [1 p] to very severe [4 p]); and distress or bother (from not at all [0 p] to very much [4 p]). Here, higher score indicate worse symptom experience.

SECONDARY OUTCOMES:
Cognitive symptoms | At hospital discharge, an average of one week
  Level of cognitive functioning is measured with The Mini Montreal Cognitive Assessment (Mini MoCA). Mini MoCA assess memory/attention; language; orientation; and delayed recall. The score can range from 0 to 15 points. Higher scores indicate better cognitive function, and 12 points or more is considered as normal.
Posttraumatic stress symptoms | At hospital discharge, an average of one week
  Posttraumatic stress symptoms is measured with Impact of event scale-revised (IES-R), a 22-item scale measuring the presence and severity of posttraumatic stress symptoms. Each item is rated on a 5-point Likert scale ranging from 0 (not at all) to 4 (extremely). The total IES-R score range is 0-88; and higher score indicate higher symptom level.
Anxiety and depression | At hospital discharge, an average of one week
  Anxiety and depression is measured with Hospital Anxiety and Depression Scale (HADS). HADS consists of 14 items, with seven each for measuring anxiety and depression. Each item can be scored on a scale from 0 (not at all) to 3 (very much). An overall score from 0 to 21 can be calculated for each subscale with the following score breakdown: 0 - 7: Normal levels of anxiety/depression; 8-10: Borderline abnormal; and > 11: Abnormal.
Physical symptoms | At hospital discharge, an average of one week
  Activities of Daily Living is measured with Katz Index of Independence in Activities of Daily Living. Katz measures the patient's ability to perform personal activities of daily living; bathing, dressing, toileting, transferring, continence, and feeding. Each item are scored as independence (1 point) or dependence (0 point). The total score can range from 0 to 6 points; a score of 2 indicates severe functional impairment; a score of 4 indicates moderate function, and a score of 6 points indicates full physical function.
Health status | At hospital discharge, an average of one week
  Health status is measured with EQ-5D-5L. This tool assess walking, personal care, common chores, pain/ discomfort, and anxiety/ depression. Each item is rated on a 5 point Likert scale from 0 (no problem) to 5 (unable to or very strong symptoms). The total score can range from 0 to 25 points, and higher score indicates better health status.
Health-related quality of life state | At hospital discharge, an average of one week
  Health-related quality of life state is measured with the visual analog scale of the EQ-5D-5L. The scale range from 0-100, with higher scores indicating better health status.

CONTACTS AND LOCATIONS:
Overall Officials: Brita Fosser Olsen, RN,PhD, Principal Investigator — Østfold Hospital Trust Postbox 300, 1714 Grålum, Norway
Locations (2):
- Norway (2):
  - Ostfold Hospital Trust, Sarpsborg, Gralum
  - Østfold Hospital Trust, Sarpsborg, Gralum

IPD SHARING:
Plan to Share IPD: No